CLINICAL TRIAL: NCT06395324
Title: Fiber Effectively Educates & Directs the Microbiome Study
Acronym: FEEDMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2117625
Record Dates: First submitted 2024-04-15; First posted 2024-05-02 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Microbial Colonization
Keywords: Fecal microbiome; Arabinose; Fecal glycome; Fecal short chain fatty acids; Fiber; High arabinose diet
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled and will consume study provided high arabinose foods during the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre, during and post high arabinose foods intake (Experimental): All individuals will enter a lead-in period consisting of a low arabinose diet, then they will consume a high arabinose diet and then back to the low arabinose diet.
  Interventions: Other: High arabinose diet

INTERVENTIONS:
Other: High arabinose diet — Participants will consume a high arabinose diet for 18 consecutive days.

SUMMARY:
The FEEDMe Study is a single-group, open label pilot study exploring how diverse, commercially available foods rich in arabinose influence the gut microbiome in adults from diverse populations.

DETAILED DESCRIPTION:
Upon enrollment, healthy adults will enter a 15-day lead-in period during which they will refrain from consuming specific foods and collect a baseline stool sample. The intervention period will be on days 16-33 during which participants will consume study provided high-arabinose foods. The follow-up period will be on days 34-49 during which participants will no longer eat the study foods and will refrain from consuming specific foods. The total duration of the study will be approximately 7 weeks. Stool samples will be collected on 3 occasions and participants will be asked to complete questionnaires, daily stool logs, dietary intake reports, and 24-hour dietary recalls throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 18-50 years of age;
* BMI between 18.5 and 34.9 kg/m2;
* Lives within a 40-mile radius from the UC Davis campus in Davis or UCDMC in - Sacramento, CA or study personnel residences;
* Consumes food at least three times (meals/snacks) per day;
* Non-alcohol consumers or those who consume alcohol in moderation defined as having up to 1 drink per day for women and up to 2 drinks per day for men;
* Normal stool frequency defined as 3 times per week to 3 times per day;
* Has been weight-stable (has not lost or gained 10% of body weight) within the past 3 months;
* Speaks, writes, and understands English to complete study activities;
* Lives in a household whereby stool samples and study food can be reliably stored without interference from other household members (i.e., excluding individuals who reside in fraternity, sorority houses whereby freezer access is open to all members);
* Lives in a household with access to Wi-Fi and/or cellular access to enable completion of electronic questionnaires (i.e., PIP forms) on their own personal computer, cell phone, or electronic device;
* Willingness to consume study-provided foods for 18 consecutive days;
* Willingness to fill out a short online survey about the amount of each study food they consumed during the two-week intervention;
* Willingness to collect stool samples on three separate days and store them in their home freezer before they (or study personnel) transport them to UC Davis;
* Willingness to complete online weekly health questionnaires;
* Willingness to complete two online enrollment questionnaires about diet and health history;
* Willingness to complete Daily Stool Logs (7 consecutive days) at 3 separate times during the study period;
* Willingness to complete two 24-hour dietary recalls by video call with study personnel (prior to each of the 3 stool collections required for the study);
* Willingness to have four in-person visits (at their homes or on campus);
* Willingness to use their personal computer, cell phone, or electronic device to meet virtually with study personnel;
* Willingness to refrain from consuming fermented foods, or foods with probiotics or probiotic supplements and other foods listed on the study materials (confounding variables of the intestinal microbiome) during the study period;
* Willingness to refrain from consuming iron containing dietary supplements (multi-vitamin is permitted) and fiber supplements during the study period;
* Willingness to refrain from changing (starting a new or discontinuing a current) routine vitamin/mineral supplement regimen during the study period;
* Willingness to refrain from changing (starting a new or discontinuing a current) routine medication regimen during the study period;
* Willingness to refrain from consuming laxatives during the study period;
* Willingness to refrain from enrolling in other experimental trials during the study period;
* Willingness to avoid binge alcohol drinking during the study period defined by the CDC as: drinking 5 or more drinks on a single occasion for men or 4 or more drinks on a single occasion for women, generally within about 2 hours;
* Willingness to refrain from using tobacco (smoking or chewing or using E-cigarettes) or smoking, vaping or consuming cannabis or use of other illicit drugs during the study period;
* Willingness to refrain from having any non-emergency, elective surgeries including dental surgery or invasive medical procedures during the study period;
* Willingness to take a study-provided urine pregnancy test if female;
* Mid- to high-income families and low-income families based on household income or eligibility for the California Supplemental Nutrition Assistance Program (SNAP) or Special Supplemental Nutrition Program for Women, Infants, and Children (WIC).

Exclusion Criteria:

* Currently pregnant or plans to become pregnant several weeks prior to enrollment and during the study period;
* Currently lactating;
* Use of restrictive diets such as caloric restriction, intermittent fasting, keto-diet, gluten-free, grain-free, dairy-free within the past 6 months;
* Known or suspected allergy (childhood allergies pre-puberty is acceptable) to milk, egg, wheat, legumes including soybeans; peanuts, tree nuts and seeds, and any fruits and vegetables used in the study;
* Known or suspected sensitivity or intolerances to any foods and ingredients used in the study (e.g., lactose intolerance, etc.) such as milk, egg, wheat, legumes including soybeans, peanuts, tree nuts and seeds and any fruits and vegetables used in the study;
* Aversions to or avoidance in eating foods and ingredients used in the study (legumes/beans, fruits, vegetables, peanuts, tree nuts and seeds);
* History of any type of eating disorder (anorexia nervosa, bulimia, etc.);
* History of any of the following: Positive infection of HIV, AIDS, hepatitis B or C; GI tract abnormalities; Any type of bariatric surgery or other gastric surgery involving the removal of sections of the GI tract (appendectomy or hernia repairs are acceptable), or gall-bladder removal; GI-related conditions such as malabsorption disease, celiac disease, Crohn's disease, colitis, inflammatory bowel disease (IBD), irritable bowel syndrome (IBS); Cancer (history of skin cancer that is in remission is acceptable), heart, liver, lung, endocrine, or kidney diseases; Type 1 or 2 diabetes mellitus; Cushing syndrome; Primary immune deficiency or autoimmune diseases; Uncontrolled hyper or hypothyroidism; uncontrolled hypertension (controlled with medication is acceptable);
* History of stomach ulcers or diagnosis with H. pylori infection; chronic gastritis within the past 12 months;
* Gastroenteritis (caused by stomach flu or food poisoning caused by virus or bacteria) within the past 4 weeks;
* Have any medical or nutritional conditions that require iron supplementation;
* Intake of iron supplements (stand-alone doses that are not part of a multi-vitamin) within the past 4 weeks;
* Positive test for COVID-19 based on a rapid test or PCR within the past 2 weeks;
* Use of oral, intramuscular or IV antibiotics or sulfonamides within the past 3 months;
* Vaccinations received less than the past 2 weeks (may enroll two weeks following treatment with vaccinations);
* Use of biologics that suppress the immune system, i.e., Lantus, Remicade, Rituxan, Humira, Herceptin, Avastin, Lucentis, Enbrel, for 2 weeks or longer or within the past 4 weeks;
* Use of injectable (or pill) weight loss medications or biologics such as Ozempic, Wegovy, Rybelsus, etc. within the past 4 weeks;
* Surgery or an invasive medical procedure within the past 3 months;
* Plan to have any elective surgeries including dental surgery or invasive medical procedures during the study period;
* Illness (flu, cold, etc.) within the past 2 weeks (free of all illness symptoms within the past 2 weeks);
* Routine use of medications found to alter the gut microbiome such as: Tylenol, aspirin, naproxen sodium or ibuprofen (except for acute uses with sickness or injury), anticholinergic inhalers, opioids, proton pump inhibitors, gastric acid suppressors (e.g., pepcid), metformin, statins, steroids (oral-inhaler is acceptable), 6-Marcaptopurine, Azathioprine or any other immunosuppressants on a daily basis within the past 6 months;
* Plans to start or plans to have changes made to a dose (including starting or adjusting an existing dose) of selective serotonin reuptake inhibitors (SSRIs), or antipsychotics during the study period;
* Plans to start or plans to have changes made to a dietary supplement regimen (vitamins/minerals/herbal supplements) or a medication regimen during the study period;
* Persistent (lasts longer than 2 weeks and less than 4 weeks) or chronic (lasts at least 4 weeks) diarrhea (loose, watery stools three or more times a day) within the past 6 months;
* Chronic constipation (fewer than 3 stools per week, stool form that is mostly hard or lumpy and difficult stool passage (need to strain or incomplete evacuation) with the past 3 months;
* Use of probiotic supplements within the past 8 weeks;
* Individuals who use laxatives more than once per week;
* Individuals who use fiber supplements more than once per week;
* Current tobacco (smoking or chewing) or E-cigarette users or individuals who quit using less than one year before enrolling in the study;
* Frequent cannabis use (eating, smoking, or vaping) defined as greater than 4 times per week and greater than 14 times per month;
* Use of illicit drugs (cocaine, crack, heroine, unprescribed fentanyl etc.);
* Excessive alcohol drinkers: For men, heavy drinking is typically defined as consuming 15 drinks or more per week. For women, heavy drinking is typically defined as consuming 8 drinks or more per week (https://www.cdc.gov/alcohol/faqs.htm);
* Individuals who currently live or plan to live within the same household during the study period or who are in intimate relationships with current or past study participants (to avoid horizontal transfer of the gut microbiome),
* Individuals who plan to travel during the stool collections and intervention phase of the study duration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Fecal microbiome | Change from baseline to days 31 and 47
  Examine changes to the concentration and distribution of fecal microbiota in response to consuming a high arabinose diet as measured by 16s rRNA sequencing and metagenomics.
Fecal glycome | Change from baseline to days 31 and 47
  Determine changes in fecal glycome in response to consumption of a high arabinose diet as measured by metagenomic analysis and mass spectrometry.
Fecal SCFAs | Change from baseline to days 31 and 47
  Determine changes in fecal SCFAs in response to consumption of a high arabinose diet as measured by mass spectrometry.
Gastrointestinal tolerance | Change from baseline to days 31 and 47
  Assess gastrointestinal tolerance to a high arabinose diet as measured by questionnaires that ask participants to report gastrointestinal symptoms. A list of GI symptoms are listed in the weekly survey and participants will select none, mild, moderate, severe or unsure. The proportion of severe responses will be compared across the study weeks.
Stool consistency and frequency | Change from baseline to days 16-33
  Determine changes in fecal consistency and frequency in response to a high arabinose diet as measured by questionnaires that ask participants to report their number of stools per day and to rank the consistency of their stools using the Bristol Stool Scale. For seven days prior to each of the three stool collections, participants will rate their stool consistency on a scale from 1-7 and these values will be averaged and compared across the three time points (pre, during and post high arabinose diet). This scale is not continuous but rather nominal and the proportion of 4 and 5 is considered "normal" stoo consistency.
Study food acceptability | Intervention period: days 31-46
  Examine overall acceptability and sensory perceptions of high arabinose commercially available products as measured by questionnaires. Participants will rate how much they like each study food after consuming each one for the first time on a continuous scale from 0 to 100 where 0 equals did not like at all and 100 equals extremely liked. The scores will be reported for each food.
Study expansion feasibility | Study period: Days 1-49
  Evaluate the overall satisfaction of participants' experience for feedback on the study protocol and study duration. At the end of the study, participants will rate their satisfaction on a continuous scale from 0 to 100, where 0 equals not satisfied at all and 100 equals extremely satisfied.
Follow-up period evaluation | Follow-up period: days 34-49
  Evaluate if 14 days of avoiding arabinose foods is a sufficient washout period to result in changes in concentration and distribution of gut microbiota as measured by 16s rRNA sequencing and metagenomics.

SECONDARY OUTCOMES:
Fecal immune markers | Change from baseline to days 31 and 47
  Determine changes in fecal immune and inflammatory markers such as levels of immunoglobulins in response to a high arabinose diet as measured by ELISA and mass spectrometry.
Fecal metabolomics | Change from baseline to days 31 and 47
  Determine changes in fecal metabolites and organic acids in response to a high arabinose diet as measured by mass spectrometry.

OTHER OUTCOMES:
Exploratory Endpoint 2 | Study period: Days 1-49
  Determine the feasibility of executing the study design in two different populations: 1) medium and high income and 2) low-income communities at-risk for gut dysbiosis by comparing attrition rates among the two groups.
Exploratory Endpoint 1 | Study period: Days 1-49
  Determine the feasibility in adults consuming a high arabinose diet over 2.5 week period by assessing adherence to the study protocol and attrition rates.
Exploratory Endpoint 3 | Study period: Days 1-49
  Determine differences for all primary and secondary endpoints between middle/high income and low-income participants in response to a high arabinose diet by stratifying data based on these two groups.
Safety Endpoints | Study period: Days 1-49
  Determine if the study resulted in any Adverse Events and Serious Adverse Events by administering a questionnaire that asks participants to report the occurrence of any illness and health care visits for sickness. Participants complete weekly questionnaires and report if they experienced any illnesses or hospital visits. The proportion of these incidence will be reported across the three time points (pre, during and post high arabinose diet).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Smilowitz, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] So D, Whelan K, Rossi M, Morrison M, Holtmann G, Kelly JT, Shanahan ER, Staudacher HM, Campbell KL. Dietary fiber intervention on gut microbiota composition in healthy adults: a systematic review and meta-analysis. Am J Clin Nutr. 2018 Jun 1;107(6):965-983. doi: 10.1093/ajcn/nqy041. PMID 29757343
- [Background] Gill SK, Rossi M, Bajka B, Whelan K. Dietary fibre in gastrointestinal health and disease. Nat Rev Gastroenterol Hepatol. 2021 Feb;18(2):101-116. doi: 10.1038/s41575-020-00375-4. Epub 2020 Nov 18. PMID 33208922
- [Background] U.S. Department of Agriculture USDoHaHS. Dietary Guidelines for Americans, 2020-2025. 2020(9th Edition).
- [Background] Castillo JJ, Couture G, Bacalzo NP Jr, Chen Y, Chin EL, Blecksmith SE, Bouzid YY, Vainberg Y, Masarweh C, Zhou Q, Smilowitz JT, German JB, Mills DA, Lemay DG, Lebrilla CB. The Development of the Davis Food Glycopedia-A Glycan Encyclopedia of Food. Nutrients. 2022 Apr 14;14(8):1639. doi: 10.3390/nu14081639. PMID 35458202
- [Background] Delannoy-Bruno O, Desai C, Raman AS, Chen RY, Hibberd MC, Cheng J, Han N, Castillo JJ, Couture G, Lebrilla CB, Barve RA, Lombard V, Henrissat B, Leyn SA, Rodionov DA, Osterman AL, Hayashi DK, Meynier A, Vinoy S, Kirbach K, Wilmot T, Heath AC, Klein S, Barratt MJ, Gordon JI. Evaluating microbiome-directed fibre snacks in gnotobiotic mice and humans. Nature. 2021 Jul;595(7865):91-95. doi: 10.1038/s41586-021-03671-4. Epub 2021 Jun 23. PMID 34163075